CLINICAL TRIAL: NCT03539042
Title: The Epigenetics of Exercise and Physical Activity in COPD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emily S. Wan, Physician and Principal Investigator, VA Boston Healthcare System
Other Study IDs: 3013
Record Dates: First submitted 2018-05-01; First posted 2018-05-29 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Copd
Keywords: DNA methylation; Physical activity; Exercise capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and urine will be collected at 2 time points via venipuncture. Plasma and buffy coat will be extracted and stored for analysis at the conclusion of the study.
  Participation in this study will not impact the course of usual clinical care (observational study).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study seeks to examine genome-wide DNA methylation patterns associated with physical activity and exercise capacity from peripheral blood collected from participants with chronic obstructive pulmonary disease (COPD) before and after participation in a structured 9-week outpatient pulmonary rehabilitation program.

DETAILED DESCRIPTION:
Individuals who are referred to pulmonary rehabilitation IN THE COURSE OF THEIR USUAL CLINICAL CARE will be invited to participate in this observational study. Participants who enroll in the study will undergo two in-person visits, once before initiating pulmonary rehabilitation classes and once at the conclusion of pulmonary rehabilitation classes. Participation in this study will not alter the course of the participants' usual clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years
* Diagnosis of COPD (defined as an FEV1/FVC<0.7 or evidence of emphysema on radiologist's read of a chest CT obtained in the course of patient's usual care)
* Referral to and participation in the VA Boston Pulmonary Rehabilitation program

Exclusion Criteria:

* Active or unstable cardiac disease
* Inability to ambulate > 1 block
* Recent acute exacerbation of COPD (defined as new or increased dose of systemic steroids and/or antibiotics for pulmonary indications)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit from Veterans referred to the VA Boston Pulmonary Rehabilitation Program who have a confirmed diagnosis of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in DNA methylation patterns | Baseline and 3-month follow up
  Baseline patterns and changes over time after participation in exercise training

SECONDARY OUTCOMES:
Change in 6MWD | Baseline and 3-month follow up
  Change in exercise capacity (assessed as 6 minute walk distance) after exercise training in pulmonary rehabilitation
Change in average daily step count | Baseline and 3-month follow up
  Change in pedometer assessed daily step count before and after exercise training in pulmonary rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Emily S Wan, MD,MPH, Principal Investigator — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual level data will be entered into an approved research repository behind the VA firewall. Data will be shared with qualified researchers (see below)
Time Frame: 3 years
Access Criteria: Prospective researchers must complete VA-required trainings in HIPAA, information security, and CITI training.